CLINICAL TRIAL: NCT02782182
Title: Perioperative FOLFIRINOX for Patients With Resectable Pancreatic Adenocarcinoma: A Pilot Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed early due to poor accrual.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1630
Record Dates: First submitted 2016-05-16; First posted 2016-05-25 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: Pancreatic ductal adenocarcinoma; FOLFIRINOX; resectable pancreatic cancer
MeSH Terms: interventions — folfirinox; Oxaliplatin; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FOLFIRINOX+surgery (Experimental): 4 cycles of pre-operative FOLFIRINOX, followed by surgery, followed by 2 more cycles of FOLFIRINOX
  Interventions: Drug: FOLFIRINOX (oxaliplatin, leucovorin, irinotecan)

INTERVENTIONS:
Drug: FOLFIRINOX (oxaliplatin, leucovorin, irinotecan) — FOLFIRINOX administered preoperatively and postoperatively

SUMMARY:
The purpose of this study is to see whether it is possible to give 8 doses of a combination of chemotherapy called FOLFIRINOX before surgery in subjects whose pancreas cancer can be removed with surgery.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the percentage of pancreatic cancer patients able to complete the full 4 months of preoperative chemotherapy and undergo a resection.

Secondary Objectives

* To assess the percentage of patients able to complete all therapy, including preoperative chemotherapy, surgery, and postoperative therapy.
* To assess treatment-related toxicity during preoperative therapy
* To assess intra-operative and post-operative complications
* To assess the histopathologic (R0/R1) resection rate after preoperative therapy
* To determine disease free survival (DFS) for patients who undergo resection.
* To determine progression free survival (PFS) for all patients
* To determine overall survival (OS) from the date of first treatment

ELIGIBILITY:
Inclusion Criteria

1. Histologic or cytologic diagnosis of adenocarcinoma of the pancreas.
2. Resectable primary tumor of the head, body or tail of the pancreas defined per NCCN Guidelines version 2.2015:

   * No extra-pancreatic disease, aside from lymphadenopathy
   * No arterial tumor contact (celiac axis, superior mesenteric artery, or common hepatic artery)
   * No tumor contact with the superior mesenteric vein or portal vein or ≤ 180° contact without vein contour irregularity
3. Confirmation of resectability by surgical oncology consultation.
4. No previous therapy for pancreatic cancer
5. Short removable metal stents rather than plastic stents are strongly encouraged but not required for palliation of initial obstructive jaundice
6. ECOG performance status of 0 or 1 (Appendix 1)
7. Age > 18 years
8. No CVA within 6 months, no MI within 6 months
9. The effects of mFOLFIRINOX on the developing human fetus are unknown. For this reason and because chemotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Negative pregnancy test in females of reproductive age
11. Anticoagulation is permitted but patients may not be on warfarin.
12. Patients must have normal organ and marrow function as defined below:

    * absolute neutrophil count >1,500/mcL
    * platelets >100,000/mcL
    * total bilirubin < 1.5X upper limits of normal
    * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
    * creatinine within normal institutional limits OR
    * creatinine clearance >60 mL/min/ per Cockroft-Gault equation for patients with creatinine levels above institutional normal.
13. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had previous chemotherapy or radiotherapy for pancreatic adenocarcinoma prior to entering the study.
2. Pathologic subtypes other than pure adenocarcinoma; acinar cell carcinoma, squamous cell carcinoma, spindle cell carcinoma, neuroendocrine cancer, and mixed types are not eligible.
3. Patients who are receiving any investigational agents.
4. Patients with borderline resectable, locally advanced or metastatic disease.
5. History of allergic reactions attributed to 5-FU, leucovorin, irinotecan or oxaliplatin or to compounds of similar chemical or biologic composition.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active liver disease including viral or non-viral hepatitis and cirrhosis, chronic diarrhea or inflammatory disease of the colon or rectum, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study. mFOLFIRINOX is a regimen containing more than one chemotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with mFOLFIRINOX, breastfeeding should be discontinued if the mother is treated with these agents. These potential risks may also apply to other agents used in this study.
8. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with mFOLFIRINOX. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
9. Currently active second malignancy other than non-melanoma skin cancer or carcinoma in-situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy and have no evidence of recurrence for at least 5 years.
10. Pre-existing neuropathy greater than grade 1.
11. Inflammatory bowel disease that is uncontrolled or on active treatment (Crohn's disease, ulcerative colitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients able to complete 4 months of preoperative chemotherapy and undergo a resection | 4 months
  Measured by percentage of successes/failures

SECONDARY OUTCOMES:
The extent of preoperative chemotherapy, surgery, and adjuvant chemotherapy. | 6 months
  Reported as a yes/no for each element of therapy.
Presence of adverse events | 6 months
  Presence of grade 3 and 4 toxicities measured according to NCI CTCAE version 4.0.
Intraoperative and post-op complications | Within 6 weeks post surgery
  Any unexpected events as determined by surgical oncologist
R0/R1 resection rates | 6 months
  Measured as proportion of patients with microscopic negative and microscopic residual tumor margin
Disease free survival | Up to 5 years
  Defined by date from surgical resection to radiographic recurrence or death
Progression free survival | Up to 5 years
  Defined by radiographic progression by RECIST criteria or death
Overall survival | Up to 5 years
  Defined by date from Cycle 1 Day 1 of preoperative chemotherapy to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States